CLINICAL TRIAL: NCT01988753
Title: Utility of Shearwave Elastography (SWE) and Non-Invasive Serum Biomarkers to Detect Fibrosis in Pediatric Patients With Liver Diseases
Brief Title: Non-invasive Biomarkers of Fibrosis in Pediatric Liver Diseases
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Daniel Leung, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-30472
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Viral Hepatitis; Liver Fibrosis; Liver Disease; Hepatitis B; Hepatitis C
Keywords: Serum Biomarkers; Sheer-wave Elastography; Ultrasound imaging; Viral hepatitis; Liver Fibrosis; Liver disease; Hepatitis B; Hepatitis C
MeSH Terms: conditions — Liver Cirrhosis; Liver Diseases; Hepatitis B; Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Shearwave elastography is a non-invasive procedure to measurement liver tissue elasticity. Images will be obtained in the right lobe of the liver through intercostal spaces with the subject lying supine with right arm abduction. A total of 10 measurements will be obtained across the liver to obtain a more comprehensive evaluation.
  2. Biomarker Analysis
  A. Blood: Blood will be drawn at the same time the IV is placed for the liver biopsy for the purposes of the serum biomarker study. If subjects return for an additional liver biopsy in the future or a standard of care visit they may be asked to provide an additional sample for biomarker analysis. Blood will be processed, aliquoted and stored by pathology.
  B. Tissue: Unstained slides from pathology will be prepared from leftover tissue taken during the liver biopsy to be stained for additional biomarker analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with Liver Fibrosis: 1. Shearwave elastography is a non-invasive procedure for assessing liver status. Measurements of liver tissue elasticity will be obtained in the right lobe of the liver by using a curvilinear transducer (C5-1, Philips Healthcare) through intercostal spaces.
  2. Biomarker Analysis
  A. Blood: Blood will be drawn at the same time the IV is placed for the liver biopsy for the purposes of the serum biomarker study. If subjects return for an additional liver biopsy in the future or a standard of care visit they may be asked to provide an additional sample for biomarker analysis. Blood will be processed, aliquoted and stored by pathology.
  B. Tissue: Unstained slides from pathology will be prepared from leftover tissue taken during the liver biopsy to be stained for additional biomarker analysis.

SUMMARY:
This study is being conducted to develop new techniques for early diagnosis of liver disease. These techniques are: Shearwave Elastography (SWE) ultrasound and blood biomarkers.

SWE ultrasound uses high-frequency sound waves to view soft tissues such as muscles and internal organs and measure stiffness. An ultrasound creates computer images that show internal body organs, such as the liver or kidneys, more clearly than regular x-ray images.

Biomarkers are biological molecules found in the blood that provide important information about liver disease.

DETAILED DESCRIPTION:
Abnormal liver biochemical and function tests are frequently detected in symptomatic patients since many screening blood test panels routinely include them. A population-based survey in the United States conducted between 1999 and 2002 estimated that an abnormal alanine aminotransferase (ALT) was present in 8.9 percent of respondents. These patients are often referred to hepatology to elucidate the cause of these abnormal liver tests and potential liver disease. Identifying the cause of specific pediatric liver diseases is critical to the management and treatment. Liver biopsy provides histological information often needed to make a conclusive diagnosis and has historically been accepted as the best way to measure liver fibrosis.

Given that the current gold standard for assessing for liver fibrosis is via liver biopsy, there are several reasons why the field is looking for a non-invasive method that correlates highly with liver histology. Hemorrhage, infection, the need to often be observed overnight, anxiety, and need for sedation are the accepted risks for all liver biopsies. The histologic grade on liver biopsy (grades 0-4) is used to grade the severity of hepatic fibrosis and make clinical decisions such as initiating treatment with antiviral or immunomodulator therapy.

Ultrasound imaging (sonography) uses high-frequency sound waves to view soft tissues such as muscles and internal organs, limited primarily by non-sound transmitting tissues such as air and bone. Ultrasound is an excellent modality for the pediatric population and provides far ranging diagnostic possibilities, limiting the use of radiation whenever possible. Sheerwave elastography is a complimentary noninvasive, real-time sonographic technique that has been shown to have a wide range of clinical applications, including the ability to assess the degree of liver fibrosis in chronic liver disease. Tissue has an inherent elasticity which may be altered by pathologic processes such as inflammation, fibrosis, and tumors. Elastography has been used extensively in breast imaging showing much promise in detecting non-compressible masses associated with an increased risk of malignancy. Elastography has the ability to assess small changes in pliability of liver tissue across the entire liver. Elasticity of tissue in the context of elastography is the ratio of tension (stress) needed to produce a relative change in length (strain), and quantifies how much pressure must be placed on tissue in order to cause elastic deformation. Ultrasonic elastography has been performed to detect hepatic fibrosis in patients with fatty liver disease in adults, but not yet in children with viral hepatitis B or C.

Performance compression ultrasound require no more than 5-10 additional minutes of imaging and have no known associated risks.

Serum fibrosis markers are promising non-invasive indicators of fibrosis and progression to cirrhosis in adult liver diseases: e.g. the commercially available Fibrotest® is used to detect hepatic fibrosis in hepatitis C and in non-alcoholic fatty liver disease (NAFLD). However, marker patterns appear to be disease and development (age) specific, making some of the adult markers of doubtful value in children. As proof of principle, in a biopsy study of another pediatric fibrosing liver entity, cystic fibrosis liver disease, specific marker patterns derived from mechanistic studies were found to highly correlate with F3/4 fibrosis vs F0/1.

The rapid onset of liver disease in some children (i.e. HBV, genotype C) indicates a need to identify early markers of liver fibrosis to help facilitate early intervention. Serum chemistries used to assess hepatic inflammation and injury are not reliable. Empirically identified markers identified by genomic, proteomic, and metabolomic technologies, as well as targeted serum marker analysis, offer new strategies with which to diagnose and predict outcomes in pediatric liver diseases. Preliminary studies in children with fibrotic liver diseases have identified specific markers reflecting matrix re-modeling, hepatic stellate cell activation and chemoattractant expression in this age group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or established liver disease
* Scheduled to have a clinically indicated liver biopsy
* Between the ages 0-17

Exclusion Criteria:

* N/A

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children will be recruited from the >2500 inpatient/outpatient referrals made to the Texas Children's Liver Center per year. We will test the utility of putative serum markers of fibrosis and fibrogenesis, obtained from patients for diagnosis and prediction of the likelihood of progression to fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Non-invasive shearwave elastography (SWE) for detecting fibrosis in children with liver disease | One year
  Philips shearwave ultrasound elastography is a non-invasive procedure for assessing liver status. It provides a virtual biopsy by using liver stiffness data to detect fibrotic changes. It turns an invasive, painful, and expensive procedure into a simple, painless one, making it easier to monitor the 30 patients and leading to a more definitive diagnosis. A commercial US scanner (iU22, Philips Healthcare) was modified to produce shearwaves and track them.

SECONDARY OUTCOMES:
Serum Biomarker analysis | One year
  Blood will be drawn at the same time the IV is placed for each of the patients the liver biopsy for the purposes of the serum biomarker study. We will study hyaluronic acid, tissue inhibitor of metalloprotease 1, collagen type IV, prolyl hydroxylase and collagen type VI due to previous reports of their biological association with advanced liver disease. Furthermore, we propose to examine the utility of putative serum markers of fibrogenesis in staging hepatic fibrosis and severity of clinical disease in pediatric viral hepatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Leung, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No